CLINICAL TRIAL: NCT01074138
Title: A Phase II, Open-Label, Single-Arm Study Evaluating the Safety, Efficacy and Pharmacokinetics of KX2-391 in Patients With Bone-Metastatic, Castration-Resistant Prostate Cancer Who Have Not Had Prior Chemotherapy
Brief Title: Safety and Efficacy Study of KX2-391 for Treatment of Bone-Metastatic, Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KXO1-002-09
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Bone-Metastatic, Castration-Resistant Prostate Cancer
Keywords: CPRC
MeSH Terms: interventions — tirbanibulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Subjects will be enrolled into a 28-day dose-escalation study. If no DLT's are observed during the first 28 days, subjects are eligible to continue treatment in the Extension Phase and can remain on treatment until toxicity occurs or until disease progression.
  Interventions: Drug: KX2-391

INTERVENTIONS:
Drug: KX2-391 — KX2-391 will be administered as a 40 mg oral dosing solution, twice daily, for 6 28-day cycles.
  Other Names: KXO1

SUMMARY:
The standard of care for patients with bone-metastatic, castrate-resistant prostate cancer is chemotherapy. If a patient elects not to choose chemotherapy, 70% will progress within 6 months. KX2-391 given orally twice a day for 6 months will be evaluated for its ability to delay/prevent disease progression in patients who have not had prior chemotherapy.

DETAILED DESCRIPTION:
This is a multi-center, single-arm, open-label, prospective phase II clinical trial evaluating the efficacy, safety and pharmacokinetics of orally administered KX2-391 in adult male patients with progressive bone-metastatic CRPC. Patients must have 1) documented bone-metastatic prostate cancer, 2) castrate levels of testosterone, 3) not received prior chemotherapy, and 4) documented disease progression based on rising PSA, progressive measurable visceral disease and/or progressive bone lesions (one criteria is sufficient) as per the Prostate Cancer Clinical Trials Working Group (PCWG2) guidelines (Scher et al 2008).

ELIGIBILITY:
Inclusion Criteria:

* The patient must provide signed informed consent prior to performing any study-related procedures;
* The patient must have histologically or cytologically confirmed prostate adenocarcinoma;
* The patient must have presence of at least one documented osseous metastasis on bone scan;
* The patient must have a castrate testosterone level <50ng/dl within 4 weeks prior to initiation of KX2-391 treatment. If chemically castrate, the patient must also agree to stay on luteinizing hormone releasing hormone (LHRH) agonist medication for the duration of the study;
* The patient must have documented disease progression as evidenced by one or more of the following 3 criteria:
* Rising PSA, defined as three rising PSA values ≥ 2 weeks apart with the 3rd value 2ng/ml or greater (historical values may be used). Rising PSA must be seen in the 3rd value relative to the 2nd value AND in the 2nd value relative to the 1st value (i.e. two consecutive rises over time muse be noted). Given potential for fluctuations in PSA values, one drop in rising PSA values over time may be seen when determining eligibility. Pre-therapy PSA doubling time may also be calculated (if there are 3 or more values 4 or more weeks apart.
* Evidence of nodal or visceral progression. Progression must be evident within 3 months prior to study entry.
* Radiographic documentation of disease is required by CT (or MRI, when CT is not available)(using RECIST 1.1 criteria) within 4 weeks of study entry.The patient must have at least 1 unidimensionally measurable lesion ≥ 20mm by conventional techniques (i.e., conventional CT or chest x-ray) OR ≥ 10mm by spiral CT scan.Only lymph nodes ≥ 20mm in diameter may be counted.CT is preferred over MRI. The radiographic measurement technique used at Baseline must be serially used throughout the duration of the study.
* Evidence of progression of bone metastases on bone scan. Appearance of ≥ 2 new lesions since the prior scan (prior scan obtained within 3 months of study entry).Documentation of bone metastases by bone scintigraphy (using PCWG2 criteria) within 4 weeks of study entry.
* The patient must have no known brain metastases (confirmation by CT and/or MRI is not required);
* The patient be a ≥ 18 year old male at the time of enrollment;
* The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2;
* The patient must have an estimated life expectancy of ≥ 6 months;
* The patient must have adequate hematopoietic function as demonstrated by 1) hemoglobin of ≥ 9.0g/dL, 2) platelet count ≥ 100,000ul, 3) WBC count ≥ x109/L, and 4) ANC ≥ 1.5 x109/L;
* The patient must have adequate hepatobiliary function as demonstrated by 1) a bilirubin level ≤ 1.5 times the upper limit of normal (ULN), unless the patient has Gilbert's syndrome in which case he/she must have a bilirubin level ≤ 2.5 times the upper limit of normal and 2) aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times the ULN;
* The patient must have adequate renal function as demonstrated by a creatinine level ≤ 1.5 times the ULN and a creatinine clearance (measured or calculated) ≥ 35 mL/min;
* Patients with partners of child-bearing potential must be willing to abstain from sexual activity or practice physical barrier contraception during study participation and for at least 3 months after completion of KX2-391 treatment;
* The patient must be able to self-administer KX2-391 and agree to adhere to the study visit schedule; study treatment schedule and other protocol requirements.

Exclusion Criteria:

* The patient has had other prior malignancy (with the exception of basal cell or squamous cell carcinoma of the skin and superficial transitional cell carcinoma of the bladder) within 3 years of study entry;
* The patient has a history of major cardiovascular or neurologic disease within the 6 months prior to enrollment, including, but not limited to, uncontrolled hypertension (at the discretion of the Investigator)< NYHA Class III or IV congestive heart failure, myocardial infarction, confirmed significant cardiac conduction abnormalities (including QTc > 0.45 sec) or arrhythmias, cerebrovascular accident(s), transient ischemic attack(s), clinically significant peripheral artery disease (i.e., claudication on walking less than one block), or other major arterial thrombotic events (e.g., pulmonary embolism) (Note: Patients with deep venous thrombosis are eligible for inclusion if they have been on a stable dose of anticoagulation therapy for at least 4 weeks prior to study entry;
* The patient has peripheral neuropathy ≥ grade 2 as defined using Common Terminology Criteria for Adverse Events (CTCAE);
* The patient has uncontrolled diabetes mellitus in the opinion of the Investigator;
* The patient has experienced hemoptysis or significant bleeding episode within 6 months prior to enrollment;
* The patient has had upper or lower gastrointestinal (GI) bleeding within 6 months prior to enrollment;
* The patient has had a GI perforation within 12 months prior to enrollment;
* The patient has had major surgery of the GI tract or a history of inflammatory bowel disease, malabsorption syndrome or other medical condition that would interfere with oral drug absorption;
* The patient has a serious or non-healing wound or ulcer;
* The patient has a known history of pathological bone fracture;
* The patient has a known history of hepatitis B, C, or human immunodeficiency virus (HIV) infection;
* The patient received moderate or strong CYP450 3A4 modulators (inducers or inhibitors) within 2 weeks or 5 half-lives (whichever is shorter) prior to initiation of KX2-391 dosing and during the study;
* The patient received prior treatment with estramustine or suramin;
* The patient received treatment with flutamide, bicalutamide, nilutamide, or ketoconazole within 4 weeks of study entry;
* The patient received prior chemotherapy for prostate cancer;
* The patient received 5α-reductase inhibitors (e.g., finasteride, dutasteride) within 4 weeks of study entry;
* The patient received other hormonal therapy [e.g., aminoglutethimide, megestrol, diethylstilbestrol (DES)] within 6 weeks of study entry;
* The patient is on other concurrent endocrine therapy, the exception of 1) steroids for adrenal insufficiency or autoimmune disease, if on a stable dose for > 3 months, 2) intermittent dexamethasone as an antiemetic (to be avoided, if at all possible); and 3) hormones for non-disease-related illnesses (e.g. insulin for diabetes);
* The patient received strontium chloride (Sr89) or samarium (Sm153) lexidronam pentasodium therapy within 12 weeks of study entry;
* The patient received extensive radiation therapy (including sternum, pelvis, scapulae, vertebrae or skull) within 4 weeks of study entry;
* The patient received extensive radiation therapy > 4 weeks before study entry and has not recovered from side effects of therapy;
* The patient received palliative low dose radiation therapy limited to the limbs within 2 weeks of initiating KX2-391;
* The patient is on bisphosphonates and the dose has changed in the 4 weeks prior to study entry (initiation of bisphosphonates during the study is not permitted);
* The patient is receiving full-dose anticoagulation therapy and dose has been modified in the 4 weeks prior to study entry (patients on low molecular weight heparin or aspirin are eligible for study enrollment);
* PT or INR is > 1.5 times the upper limit of normal and the patient is not on any anti-coagulation therapy or anti-platelet agents;
* The patient is expected to initiate chemotherapy or palliative radiotherapy while on the study;
* The patient is either currently receiving or is expected to receive treatment with filgrastim (G-CSF), pegfilgrastim, or sargramostim (GM-CSF) during the study period (these medications and therapies may only be initiated when clinically indicated during the study);
* The patient has had major surgery within 4 weeks of study entry;
* The patient has had major surgery within > 4 weeks prior to study entry and has not fully recovered from the surgery;
* The patient received other investigational agents/therapies within 28 days of study entry;
* The patient has persistent ≥ grade 2 treatment-related toxicity from prior anti-cancer therapy, including other investigational agents;
* The patient has any other medical condition or serious intercurrent illness that, in the opinion of the Investigator, may make it undesirable for the patient to participate in the study, including, but not limited to, end organ failure, coagulation disorder, hemolytic condition (e.g. sickle cell disease) or active infection;
* The patient has any other condition(s) which could significantly interfere with protocol compliance, including, but not limited to, dementia, psychosis, cognitive impairment, or other major psychiatric disorder;
* The patient has previously participated in the Phase I clinical trial of KX2-391.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who do not have clinical or radiographic progression | 24 weeks
  At screening/baseline, target lesions will be identified and measured by CT scan and bone lesions will be enumerated by bone scintigraphy. At 12 and 24 weeks after treatment with KX2-391, patients will be assessed by CT and bone scan to assess whether radiographic progression has occurred. At monthly visits and throughout the study, clinical progression will be evaluated.

SECONDARY OUTCOMES:
Determine the proportion of patients who do not have PSA progression | 24 weeks
  PSA will be measure at baseline and at the start of each of 6, 28 day cycles
Determine the pharmacokinetics of KX2-391 | 24 weeks
  Pharmacokinetic parameters will be determined in patients receiving 40 mg KX2-391, twice daily.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Carducci, MD, Principal Investigator — Johns Hopkins University; Min-Fun Rudolf Kwan, MD, Study Director — Kinex Pharmaceuticals
Locations (5):
- United States (5):
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Wayne State University-Karmanos Cancer Center, Detroit, Michigan
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Scher HI, Halabi S, Tannock I, Morris M, Sternberg CN, Carducci MA, Eisenberger MA, Higano C, Bubley GJ, Dreicer R, Petrylak D, Kantoff P, Basch E, Kelly WK, Figg WD, Small EJ, Beer TM, Wilding G, Martin A, Hussain M; Prostate Cancer Clinical Trials Working Group. Design and end points of clinical trials for patients with progressive prostate cancer and castrate levels of testosterone: recommendations of the Prostate Cancer Clinical Trials Working Group. J Clin Oncol. 2008 Mar 1;26(7):1148-59. doi: 10.1200/JCO.2007.12.4487. PMID 18309951
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774